CLINICAL TRIAL: NCT04534244
Title: Management of Tributary Veins in Superficial Venous Insufficiency of the Lower Limbs: Impact of Endovenous Steam Treatment Versus Phlebectomy on Quality of Life
Brief Title: Impact of Endovenous Water Vapor Treatment on Quality of Life in Superficial Venous Insufficiency of the Lower Limbs
Acronym: INVOLVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The medical device is no longer available for the clinical trial
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: API/2020/103
Record Dates: First submitted 2020-08-04; First posted 2020-09-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-05

CONDITIONS: Venous Insufficiency of Leg

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Treatment of the tributary veins by phlebectomy
- Experimental group (Experimental): Endovenous steam treatment of the tributary veins
  Interventions: Device: VBox Hybrid

INTERVENTIONS:
Device: VBox Hybrid — Medical device intended to treat permanent venous insufficiency of saphenous veins and tributary veins in patients with superficial venous reflux
  Arms: Experimental group

SUMMARY:
The prevalence of superficial chronic venous insufficiency (CVI) of the lower limbs is estimated at 18 million French people. The number of patients operated for varicose veins is around 300,000 per year. Post-operative complications such as venous ulcer, venous thrombosis and varicose vein rupture require a lot of medical care. Varicose veins are responsible for a decrease in quality of life and represents 1 to 2% of total health expenditure.

Currently, operating techniques tend towards minimally invasive procedures in order to minimize the surgical trauma, improve patient comfort and reduce the time of postoperative work stoppages.

This study aims to compare two surgical techniques for the treatment of superficial chronic venous insufficiency of the lower limbs : phlebectomy, the gold-standard technique, and endovenous steam treatment. Several studies have already been carried out on endovenous steam treatment for saphenous veins but none has been published concerning the tributary veins.The main objective of INVOLVE is to assess the quality of life of patients 1 month after surgery. Clinical improvement and economic impact will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been menopausal for at least 24 months, surgically sterilized, or, for women of childbearing potential, use an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, double-barrier method, contraceptive patches)
* Signature of the informed consent to participate indicating that the subject has understood the purpose and procedures required by the study and that he agrees to participate in the study and to comply with the requirements and restrictions inherent in this study
* Affiliation to a French social security scheme or beneficiary of such a scheme
* Patient with a reflux of the tributary veins, associated or not with a reflux of the large saphenous veins
* Patient with a reflux of the tributary veins already treated for a reflux at the saphenous level
* Clinical stage between C2 and C5 (from the CEAP classification). Diameter of the vein between 3 and 13 mm
* Patient treated with one or two lower limbs
* Patient able to understand and complete a quality of life questionnaire

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and / or weak cooperation anticipated by the investigator
* Subject without health insurance
* Pregnant woman
* Subject in the period of exclusion from another study or provided for by the "national file of volunteers"
* Patient with an absolute or relative contraindication to the treatment of his varicose veins by an endovenous technique
* Venous insufficiency at the expense of the small saphenous vein
* Patient with a history of venous thrombosis
* Patient with hemostasis disorders
* Patient with an associated severe pathology (cancer, heart failure, renal failure)
* Patient treated with sclerotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of the quality of life relative to the health of patients after endovenous steam treatment versus phlebectomy of the tributary veins | one month after the intervention
  Questionnaire : VEnous INsufficiency Epidemiological and Economic Study on Quality of Life/Symptoms (VEINES-QOL/Sym) : target dimension " VEINES-QoL symptom summary score ". High values indicate better outcomes.

SECONDARY OUTCOMES:
Comparison of the evolution of the quality of life relating to health of patients after endovenous steam treatment versus phlebectomy of the tributary veins | 8-15 days, 3, 6, 9 and 12 months after the intervention
  Questionnaires : VEnous INsufficiency Epidemiological and Economic Study on Quality of Life/Symptoms (VEINES-QOL/Sym), 36-Item Short Form Survey Instrument (SF36).
  The scores range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Comparison of occlusion of the tributary veins after endovenous steam treatment versus phlebectomy of the tributary veins | 8-15 days and one year after the intervention
  Occlusion rate evaluated by Doppler ultrasound
Evaluation of the period of resumption of activity for people in activity after endovenous steam treatment versus phlebectomy of the tributary veins | up to 1 year
  Duration of work stoppage for working people

OTHER OUTCOMES:
Comparison of secondary complications after endovenous steam treatment versus phlebectomy of the tributary veins | 8-15 days, 1, 6 and 12 months after the intervention
  The frequency, nature and severity of adverse events or immediate complications: hematomas, infections and burns requiring or not requiring intervention
Comparison of postoperative pain after endovenous steam treatment versus phlebectomy of the tributary veins | Daily for the first 8 days after surgery
  Assessment of daily pain by the visual analogue pain assessment scale for 8 days. The scores range from zero where the respondent has the most pain to 10 where the respondent has the least pain.
Comparison of the clinical improvement felt by the patient | 1, 6 months and one year after the intervention
  Clinical improvement felt by the patient assessed by the Venous Clinical Severity Score (VCSS).
  Scores that can be obtained range between 0 and 30. Low values indicate better outcomes.
Evaluation of the economic impact of endovenous steam treatment in the management of superficial venous insufficiency of the lower limbs (cost-utility and cost-effectiveness analyzes) | 8-15 days, 1, 3, 6, 9 and 12 months after the intervention
  Estimation of the differential cost-result ratio, evaluation of utility via EQ-5D Low values indicate better outcomes